CLINICAL TRIAL: NCT04452994
Title: Individual Patient IND Expanded Access Program JNJ-68284528, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy for Patient J.M. With Multiple Myeloma
Brief Title: Individual Patient Investigational New Drug (IND) Expanded Access Program of JNJ-68284528, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy for Participant With Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108848
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: JNJ-68284528 — JNJ-68284528 will be administered as a single intravenous (IV). The target dose will be the recommended Phase 2 dose (RP2D) of 0.75*10^6 chimeric antigen receptor (CAR)-positive viable T cells per kilogram (cells/kg) (range: 0.5 to 1.0*10^6 CAR-positive viable T cells/kg).

SUMMARY:
The purpose of this individual-patient investigational new drug (IND) single patient request (SPR) is to provide participants treatment with JNJ-68284528, an investigational product prior to its marketing authorization. Such access may be considered for participants with serious/life-threatening diseases or conditions, where there exists no alternative treatments or where alternative treatments have been exhausted.

Age Groups: Child, Adult, Older Adult